CLINICAL TRIAL: NCT04025801
Title: Heidelberg Retina Tomograph (HRT) in Vivo Confocal Microscopy to Evaluate the Ocular Surface Disorders of Healthy and Diseased Individuals
Brief Title: Heidelberg In Vivo Confocal Microscopy to Evaluate the Ocular Surface Disorders of Healthy and Diseased Individuals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201903090RINB
Record Dates: First submitted 2019-07-02; First posted 2019-07-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: Healthy Individuals; Diabetes; Hypertension; Fabry Disease; Metabolic Disease; Alzheimer Disease; Dementia; Limbal Insufficiency; Phlyctenulosis; Ocular Rosacea; Graft Versus Host Disease in Eye; Dry Eye Syndrome
Keywords: confocal microscopy,cornea
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Fabry Disease; Metabolic Diseases; Alzheimer Disease; Dementia; Rosacea; Dry Eye Syndromes; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In vivo confocal microscopy (IVCM) has been used in clinical settings for more than 25 years, and is noninvasive, rapid and easily repeatable technique to investigate ocular surface disorders. It enables morphological and quantitative analysis of ocular surface microstructure. [1-3] As the technology advances, new IVCM machine, Heidelberg Retinal Tomograph with Rostock Corneal Module (HRT-RCM), was developed. Hardware and software modifications and acquisition techniques continue to expand the applications of the HRT-RCM for quantitative in vivo corneal imaging at the cellular level. The new software can access the corneal nerve more accurate. Here the investigators proposed this Institutional Review Board (IRB) to collect healthy persons and cases of different systematic diseases as well as etiologies of ocular surface diseases.

DETAILED DESCRIPTION:
Heidelberg Retina Tomograph (HRT) in vivo Confocal Microscopy to Evaluate the Ocular Surface Disorders of Healthy and Diseased Individuals

The purpose of this study is to evaluate the cornea of healthy persons and cases of differ-ent systematic diseases as well as etiologies of ocular surface diseases.

1. In vivo confocal microscopy (IVCM)

Three main confocal systems have been developed for IVCM:

1. the Tandem Scanning Confocal Microscope (TSCM) [4-6]
2. the ConfoScan 4 (Nidek Technologies Srl, Padova, Italy) [7-8]
3. the Heidelberg Retinal Tomograph with Rostock Corneal Module (HRT-RCM, Heidelberg Engineering, Ges.m.b.H., Dossenheim, Germany [9-10] The HRT-RCM is a laser scanning confocal microscope, operating by scanning a 670 nm laser beam in a raster pattern over the field of view. The system uses a high numerical aper-ture 63x objective lens (0.9 NA), and produces images with high contrast and better axial resolution (7.6 µm) than other in vivo confocal systems (9 µm for the TSCM and 24 µm for the ConfoScan). The HRT-RCM provides new built-in software for 3D imaging of the corneal structure.

Quantitative imaging of the subbasal nerve plexus could be performed by CCMetrics sys-tem, a custom software program developed at the University of Manchester. [11-12] The IVCM has the advantage of imaging through moderately opaque tissues (scarring or edema of the cornea) and also observes the dynamic process in the cornea, i.e. inflammatory reaction monitoring in infectious keratitis, wound healing after refractive surgery.[13-14]

The use of IVCM in the scientific research has been expanding rapidly over the past years. It has also been implemented for the clinical diagnosis of different ocular surface conditions as well as screening tool for patients undergoing treatment. The following are indication of IVCM:

1. Normal central cornea (aging, contact lens wear-related changes)
2. Dry eye disease
3. Corneal ectatic disorders, dystrophies, degenerations
4. Iridocorneal endothelial syndrome (ICE) syndromes
5. Keratitis (microbial, fungal, parasitic, viral)
6. Post-surgical evaluation of the cornea (cataract surgery, Laser ASsisted In situ Keratomileusis-LASIK, Laser Epithelial Keratomileusis-LASEK, Photorefractive keratectomy, keratoplasty)
7. Corneal deposits (pseudoexfoliation syndrome, drug-induced )
8. Systemic diseases (DM, Parkinson's disease, systemic lupus erythematosus, Rheumatoid arthritis, Alzheimer's disease and dementia)
9. Evaluation of the conjunctiva ( conjunctivitis, neoplasia )
10. Limbal stem cell deficiency ( chemical or thermal injury, Stevens-Johnson syndrome )

Study procedures Before examination, each patient signs the written informed consent. The patients undergo HRT in vivo confocal microscopy. Theses exam will be repeated every 3-6 months according to the disease status. In vivo confocal microscopy is routinely used examination modality for ocular surface disorders.

(1) In vivo confocal microscopy In vivo confocal microscopy was performed with the HRT in vivo confocal microscopy real-time confocal microscope (Heidelberg Engineering, Ges.m.b.H., Dossenheim, Germany) . Its auto-scan software provides the automatic alignment and recording. The results would be analyzed using CCMetrics system, a custom software program developed at the University of Manchester.

Before examination, one drop of topical anesthetic solution (proparacaine 0.5%, Alcaine) was instilled onto the ocular surface. After proper preparation, one drop of Vidisic gel (Bausch & Lomb, Ges.m.b.H., Berlin, Germany) was applied. The patients were instructed to gaze in the direction opposite to the region of measurement. The scanning was performed continuously from the superficial conjunctiva to the stromal layer

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 20 years; patient or the legal representative is able to read and sign an informed consent form.
* Patient with clear conscious and can follow the instruction of opening eyes and movement toward all direction.
* Patient with one of the diagnosis listed below:

  1. healthy individuals
  2. patient with systematic diseases: diabetes, hypertension, Fabry disease, metabolic diseases, Alzheimer's disease and dementia [15]…etc.
  3. patient with ocular surface problems: a. limbal insufficiency b. phlyctenulosis c. ocular rosacea e. ocular graft-versus-host disease (GVHD) f. dry eye syndrome (both aqueous deficiency or increased evaporative forms of dry eyes) h. after corneal transplantation i. other ocular surface diseases (long term use of anti-glaucoma eye drops)

Exclusion Criteria

1. Age < 20-year-old.
2. Pregnancy.
3. Cannot cooperate with confocal microscopy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hospital patients and healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Confocal microscopy exam of sub-basal corneal nerve fibre density (NFD) by using the CCMetrics software | Baseline, 3 months and 6 months.
  After corneal confocal microscopy exam, we will obtain outcome measures by using the CCMetrics software:
  Nerve fibre density (NFD) which is defined as the number of main nerves/frame. In healthy group, the measurements will be once. In the patient, the measurements will be every 3 or 6 months.
  The change of NFD will be documented and compared.
Confocal microscopy exam of sub-basal corneal nerve branch density (NBD) by using the CCMetrics software | Baseline, 3 months and 6 months.
  After corneal confocal microscopy exam, we will obtain outcome measures by using the CCMetrics software:
  Nerve branch density (NBD) number of main branches/frame. In healthy group, the measurements will be once. In the patient, the measurements will be every 3 or 6 months.
  The change of NBD will be documented and compared.
Confocal microscopy exam of sub-basal corneal nerve fibre length (NFL) by using the CCMetrics software | Baseline, 3 months and 6 months.
  After corneal confocal microscopy exam, we will obtain outcome measures by using the CCMetrics software:
  Nerve fibre length (NFL) which is the total length of all nerves/frame. In healthy group, the measurements will be once. In the patient, the measurements will be every 3 or 6 months.
  The change of NFL will be documented and compared.
Confocal microscopy exam of sub-basal corneal nerve fibre tortuosity (NFT) by using the CCMetrics software | Baseline, 3 months and 6 months.
  After corneal confocal microscopy exam, we will obtain outcome measures by using the CCMetrics software:
  Nerve fibre tortuosity (NFT) of the main nerves/frame. In healthy group, the measurements will be once. In the patient, the measurements will be every 3 or 6 months.
  The change of NFT will be documented and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan